CLINICAL TRIAL: NCT03261986
Title: A Prospective RSA and Clinical Evaluation of the Trident II Acetabular Cup
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Midwest Orthopaedics at Rush (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-066
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Total Hip Arthroplasty; Acetabular Cup
Keywords: Trident; RSA; THA
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Trident II acetabular cup (Other): Subjects receive the Trident II acetabular cup and RSA beads and undergo a series of post-operative RSA exams.
  Interventions: Radiation: Radiostereometric Analysis; Procedure: total hip arthroplasty with RSA bead implantation

INTERVENTIONS:
Radiation: Radiostereometric Analysis — RSA exams of the operative hip are received post-op day 1, and at 6 weeks, 3 months, 6 months, 1 year and 2 years following surgery
Procedure: total hip arthroplasty with RSA bead implantation — Patients receive RSA beads inserted into the bone surrounding the Trident II implant.

SUMMARY:
The objective of this study is to use radiostereometric analysis (RSA) and clinical outcome measures to evaluate early post-operative implant stability and the clinical performance of Stryker's Trident II Acetabular Cup.

DETAILED DESCRIPTION:
The proposed study is a prospective evaluation of data from patients undergoing primary total hip arthroplasty using the Trident II acetabular cup. Fifty patients will be recruited for this study. All patients that qualify for the study per the inclusion-exclusion criteria and provide written informed consent will receive the Trident II acetabular cup and RSA beads. Implant stability, through RSA, will be measured throughout the first two postoperative (post-op) years per the following schedule: immediate post-op and 6 weeks, 3 months, 6 months, 1 year, and 2 years following surgery. Patients will be discharged and seen for follow-up assessments as per standard of care. Adverse events that are related to the index joint will be collected. Health outcome questionnaires will be collected. The health outcome questionnaires will include: EQ-5D, HOOS JR and Harris Hip Score. Health outcome questionnaires will be completed pre-operatively and again at 6 weeks, 3 months, 6 months, 1 year and 2 years following surgery. Conventional x-ray analysis will be performed pre-operatively and again at 6 weeks, 1 year and 2 years following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic arthritis of the hip indicating surgical intervention
2. Scheduled to undergo a primary total hip arthroplasty
3. Patient is a candidate for the Trident II acetabular cup in accordance with product labeling -

Exclusion Criteria:

1. Patients less than 18 years of age, or older than 85 years of age.
2. Severe hip dysplasia (Crowe Type III or IV) in the affected hip
3. History of congenital dislocation
4. Prior arthroplasty of the affected hip
5. Active or prior infection of the affected hip
6. Morbid obesity (BMI > 40)
7. Medical condition precluding major surgery
8. Severe osteoporosis
9. Neuromuscular impairment
10. Patients with known allergy to metals
11. Pregnancy
12. Patients on dialysis or creatinine > 2.0
13. Patient is immuno-suppressed -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2020-10-09 (Estimated); Study Completion 2022-02-09 (Estimated)

PRIMARY OUTCOMES:
Does the Trident II Cup achieve acceptable fixation to the underlying bone? | 3 years
  The Trident II Cup proximal migration will be assessed. Migration of less than 0.2mm at 2 years and without continuous migration between post-operative year 1 and 2 will indicate acceptable fixation.

SECONDARY OUTCOMES:
What are the migration patterns of the Trident II acetabular cup over the first two post-operative years? | 3 years
  Migration patterns will be assessed using RSA analysis.
Is there a significant difference in health status and functional outcome before and after hip arthroplasty using Trident II Cup? | 3 years
  The health status and functional outcome will be assessed via Harris Hip Score.
Is there a significant difference in health status and functional outcome before and after hip arthroplasty using Trident II Cup? | 3 years
  The health status and functional outcome will be assessed via EQ-5D.
Is there a correlation between radiolucent lines measured by Charnley-DeLee zone analysis and migration characteristics using RSA? | 3 years
  X-ray radiographs will be taken at pre-op, 6 weeks, 1 year and 2 year appointments. It may take up to 3 years after study start for all patients to reach the 2 year visit mark, depending on how long enrollment takes.
Can inducible displacements measured at 1 year post-operative distinguish patients identified by RSA measurements as having inadequate fixation? | 2 years
  Inducible displacements will be measured using RSA exams at the 1 year follow-up. It may take up to 2 years after study start for all patients to reach the 1 year visit mark, depending on how long enrollment takes.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sporer, MD, Principal Investigator — Midwest Orthopaedics at Rush
Locations (1):
- Midwest Orthopaedics at Rush, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No